CLINICAL TRIAL: NCT05392517
Title: Effects of Self-mobilization Techniques on Pain, Range of Motion and Function in Patients With Chronic Pain
Brief Title: Effects of Self-mobilization Techniques in Chronic Thoracic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/22/0123 Ali
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Thoracic
Keywords: manual therapy; pain; Range of motion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): self-mobilization technique
  Interventions: Other: self-mobilization technique along with conventional therapy
- Group B (Other): : conventional treatment
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: self-mobilization technique along with conventional therapy — Group A will be treated with self-mobilization technique of thoracic spine with the frequency of 2 sets of 10 repetitions thrice per week for a total of six weeks and conventional treatment.
  Self-mobilization technique will be comprised of self-mobilization technique using tennis balls and foam roller. The participant will be supine with knees in 90-degree flexion.
  * Mobilization Technique 1: Cross your arms over your chest so that you are in slight flexion and then slowly begin to move your shoulders and head closer to the floor placing the mid back into extension over the balls joined to make mobilization device. Hold this position for 3 seconds and then return to the flexed position.
  * Mobilization Technique 2: Lying lengthwise on the foam roller, clasp your hands together in front of you, above your chest with arms straight. Slowly move your arms above your head until you feel a good stretch. This exercise should be pain free. Hold stretch for 30- 60 seconds.
  Arms: Group A
Other: conventional therapy — Group B will be treated with the conventional treatment (heating pad, ultrasound, thoracic strengthening exercises
  Arms: Group B

SUMMARY:
A Randomized clinical trial will be conducted at Actilife physiotherapy Rehabilitation center, Horizon Hospital Lahore through a convenient sampling technique on patients who will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with the self-mobilization technique of thoracic spine and Group B will be treated with thoracic stretching exercises at a frequency of 2 sets with 6 repetitions and thrice a week. Outcome measures will be NPRS, Goniometer, and Oswestry disability index for thoracic spine after 6 weeks. Data will be analyzed during SPSS software version 21.

DETAILED DESCRIPTION:
Chronic thoracic pain is pain that originates from the cervicothoracic junction and extends to the lower thoracic vertebrae. It is caused by strain in the thoracic spine area, sustained postures of the neck and thoracic region, sitting on the computer for a long time in slouched position, or overuse of the thoracic spine. This study aims to see the effects of the self-mobilization technique of the thoracic spine on pain, range of motion, and function in patients with chronic thoracic spine pain. A Randomized clinical trial will be conducted at Actilife physiotherapy Rehabilitation center, Horizon Hospital Lahore through a convenient sampling technique on patients who will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with the self-mobilization technique of thoracic spine and Group B will be treated with thoracic stretching exercises at a frequency of 2 sets with 6 repetitions and thrice a week. Outcome measures will be NPRS, Goniometer, and Oswestry disability index for thoracic spine after 6 weeks. Data will be analyzed during SPSS software version 21. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* chronic thoracic pain minimum 3 months

Exclusion Criteria:

* Soft tissues disease
* Bony disease
* Surgical history of thoracic spine
* Fracture history of thoracic spine
* Tumor
* Psychological disorders
* Traumatic injury

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 6th Week
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain
Universal Goniometer (UG) | 6th Week
  It will measure range of motion of thoracic spine.
Oswestry disability index | 6th Week
  It is a self-reported measurement tool that measures both pain and functional status and is used for evaluating disability caused by thoracic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil-ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Actilife physiotherapy rehabilitation centre, Horizon hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortega-Santiago R, Maestre-Lerga M, Fernandez-de-Las-Penas C, Cleland JA, Plaza-Manzano G. Widespread Pressure Pain Sensitivity and Referred Pain from Trigger Points in Patients with Upper Thoracic Spine Pain. Pain Med. 2019 Jul 1;20(7):1379-1386. doi: 10.1093/pm/pnz020. PMID 30821833
- [Background] Bikbov MM, Kazakbaeva GM, Zainullin RM, Salavatova VF, Gilmanshin TR, Arslangareeva II, Nikitin NA, Mukhamadieva SR, Yakupova DF, Panda-Jonas S, Khikmatullin RI, Aminev SK, Nuriev IF, Zaynetdinov AF, Uzianbaeva YV, Jonas JB. Prevalence of and factors associated with low Back pain, thoracic spine pain and neck pain in Bashkortostan, Russia: the Ural Eye and Medical Study. BMC Musculoskelet Disord. 2020 Feb 1;21(1):64. doi: 10.1186/s12891-020-3080-4. PMID 32007098
- [Background] Heneghan NR, Baker G, Thomas K, Falla D, Rushton A. What is the effect of prolonged sitting and physical activity on thoracic spine mobility? An observational study of young adults in a UK university setting. BMJ Open. 2018 May 5;8(5):e019371. doi: 10.1136/bmjopen-2017-019371. PMID 29730619
- [Background] de Vitta A, Campos LD, Bento TP, Felippe LA, Ramos WL, Fernandes JAA, et al. Thoracic Spine Pain in Adolescents and Its Association With Electronic Devices and Other Factors. 2020.
- [Background] Fredin K, Loras H. Manual therapy, exercise therapy or combined treatment in the management of adult neck pain - A systematic review and meta-analysis. Musculoskelet Sci Pract. 2017 Oct;31:62-71. doi: 10.1016/j.msksp.2017.07.005. Epub 2017 Jul 21. PMID 28750310
- [Background] Yamak B, İmamoğlu O, İslamoğlu İ, Çebi MJETS. The effects of exercise on body posture. 2018;13(18).
- [Background] Nakamaru K, Aizawa J, Kawarada K, Uemura Y, Koyama T, Nitta O. Immediate effects of thoracic spine self-mobilization in patients with mechanical neck pain: A randomized controlled trial. J Bodyw Mov Ther. 2019 Apr;23(2):417-424. doi: 10.1016/j.jbmt.2018.05.008. Epub 2018 Jun 1. PMID 31103129
- [Background] Puntumetakul R, Pithak R, Namwongsa S, Saiklang P, Boucaut R. The effect of massage technique plus thoracic manipulation versus thoracic manipulation on pain and neural tension in mechanical neck pain: a randomized controlled trial. J Phys Ther Sci. 2019 Feb;31(2):195-201. doi: 10.1589/jpts.31.195. Epub 2019 Feb 7. PMID 30858662
- [Background] Kim S-j, Kim S-y, Lee M-jJPTK. The Effects of Thoracic Spine Self-mobilization Exercise Using a Tool on Pain, Range of Motion, and Dysfunction of Chronic Neck Pain Patients. 2020;27(1):1-10.
- [Background] Joshi S, Balthillaya G, Neelapala YVR. Immediate effects of cervicothoracic junction mobilization versus thoracic manipulation on the range of motion and pain in mechanical neck pain with cervicothoracic junction dysfunction: a pilot randomized controlled trial. Chiropr Man Therap. 2020 Aug 7;28(1):38. doi: 10.1186/s12998-020-00327-4. PMID 32762708